CLINICAL TRIAL: NCT06570252
Title: A Randomized, Controlled, Double Blinded National Single-center Study to Evaluate the SteriwaveTM Antimicrobial Photodynamic Therapy System for Preoperative Nasal Cavity Decolonization in Adult Patients.
Brief Title: Preoperative Microbial Reduction of the Nasal Cavity With Antimicrobial Photodynamic Therapy (aPDT).
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Ondine Biomedical Inc. (Industry); University Hospital, Zürich, Innovation Pool (Unknown)
Responsible Party: Principal Investigator, Harald Essig, Prof. Dr. med. Dr. med. dent.; Clinical director a.i Department for Craniomaxillofacial Surgery, University of Zurich
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Nasal aPDT 01
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Efficacy of Preoperative Microbial Reduction in the Nasal Cavity Using Antimicrobial Photodynamic Therapy (aPDT)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group - nasal aPDT (Experimental): 1. Swabbing the formulation applicator (soft swab pre-saturated with the photosensitizer formulation) inside the patient's nostrils.
  2. Connection of the nasal light illuminator to the light source and insertion of the nasal light illuminator into the patient's right and left nostrils.
  3. Experimental group: Activation of the light source and illumination of the nose and nasopharynx for 2 minutes.
  4. Repetition of steps 1.-3. to complete photo disinfection of all nasal regions.
  Duration of study intervention: 14 minutes
  Intervention is performed during preparations prior to surgery and followed by regular disinfection of oral cavity (not nasal cavity) according to hospital standards after nasal swab test.
  Interventions: Device: activated Light Source (aPDT)
- Control Group - no light activation (Active Comparator): 1. Swabbing the formulation applicator (soft swab pre-saturated with the photosensitizer formulation) inside the patient's nostrils.
  2. Connection of the nasal light illuminator to the light source and insertion of the nasal light illuminator into the patient's right and left nostrils.
  3. no activation of light source
  4. Repetition of steps 1.-3. to complete control intervention.
  Duration of treatment: 14 minutes
  Intervention is performed during preparations prior to surgery and followed by regular disinfection of oral cavity (not nasal cavity) according to hospital standards after nasal swab test.
  Interventions: Device: non activated Light Source (Control)

INTERVENTIONS:
Device: activated Light Source (aPDT) — Application of SW3100 Formulation (0.2% chlorhexidine gluconate and methylene blue) in both nostrils followed by placing the SW3200 Nasal Light Illuminator with one channel per nostril.
  Activation of SW4000 Light Source (Class 1 Laser Device) that generates red light consisting of 2 channels of 700 mW, 664 nm light (continuous wave) used to activate the disinfecting formulation.
  Duration of illumination 2 minutes
  Other Names: SteriwaveTM Nasal Photodisinfection System; SW4000 Light Source; SW3200 Nasal Light Illuminator; SW3100 Formulation Applicator
  Arms: Experimental Group - nasal aPDT
Device: non activated Light Source (Control) — Application of SW3100 Formulation (0.2% chlorhexidine gluconate and methylene blue) in both nostrils followed by placing the SW3200 Nasal Light Illuminator with one channel per nostril.
  No activation of SW4000 Light Source
  Waiting for 2 minutes
  Other Names: SW3100 Formulation Applicator; SW3200 Nasal Light Illuminator
  Arms: Control Group - no light activation

SUMMARY:
The goal of this clinical trial is to investigate the preoperative microbial reduction of the nasal cavity using Photodynamic Therapy (aPDT) in adult patients undergoing surgical intervention at the Department for Craniomaxillofacial Surgery, University Hospital Zurich, Switzerland.

The main question the trial aims to answer is:

- Does aPDT reduce microbial colonization in the nasal cavity more effectively 5 minutes after treatment compared to the baseline (before intervention)?

Participants will be randomized into two groups:

* Study Group: Nasal cavity photodisinfection using aPDT.
* Control Group: Treatment with 0.2% chlorhexidine gluconate and non-light activated methylene blue.

Researchers will compare the effectiveness of aPDT against the control treatment in reducing microbial colonization of the nasal cavity.

Study Procedure:

1. Nasal swab for baseline microbial colonization.
2. Application of 0.2% chlorhexidine gluconate and methylene blue.
3. Insertion of nasal light illuminator into the patient's nostrils:

   * Study Group: Activation of the light source.
   * Control Group: No activation of the light source.
4. Nasal swab taken 5 minutes after the intervention to assess microbial reduction.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female ≥ 18 years of age
* surgical intervention in general anesthesia at the department of Oral and Maxillofacial Surgery of University Hospital Zurich

Exclusion Criteria:

* inability to tolerate insertion of the light illuminator or the photosensitizer applicator due to anatomic variations (size, shape of oro-nasal region) or disease
* inability to follow the procedure of the investigation, e.g., due to language problems or psychological disorders of the subject
* known allergic reactions to components of the nasal decolonization treatment, including methylene blue or chlorhexidine gluconate
* planed surgery in the nasal cavity
* necessary nasal intubation for surgical intervention
* vulnerable persons (subjects incapable of judgment or subjects under tutelage)
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Bacterial colonization 5 minutes after aPDT microbe groups, expressed as a score (range 0-27). | 5 minutes after Intervention
  Relative abundance of CFU (colony forming unit) over nine analyzed microbe groups (expressed as score (range 0-27)) adjusted to the baseline measure 3 minutes pre-intervention.
  Name CFU's Score "not detectable" below detection limit 0 "sporadic" <10^4 1 "moderate" 10^4 - 10^5 2 "plentful" >10^5 3
  Nine microbial subgroups for analysis:
  1. ß-hemolytic (group A and group B) Streptococcus
  2. Staphylococcus aureus (with discrimination in MSSA and MRSA)
  3. Coagulase negative Staphylococcus species (incl. Staphylococcus epidermidis)
  4. a-hemolytic Streptococcus species (oral or viridans-group Streptococci)
  5. Corynebacterium species
  6. Candida species
  7. Enterobacterales
  8. Actinomyces species and miscellaneous aerotolerant bacteria
  9. Anaerobic bacteria with focus on Propionibacterium

SECONDARY OUTCOMES:
Bacterial colonization 14 (+/-1) days after aPDT | 14 (+/- 1) days
  Bacterial colonization 14 (+/-1) days after aPDT across the nine analyzed microbe groups and expressed as score (range 0-27).
  Name CFU's Score "not detectable" below detection limit 0 "sporadic" <10^4 1 "moderate" 10^4 - 10^5 2 "plentful" >10^5 3
  Nine microbial subgroups for analysis:
  1. ß-hemolytic (group A and group B) Streptococcus
  2. Staphylococcus aureus (with discrimination in MSSA and MRSA)
  3. Coagulase negative Staphylococcus species (incl. Staphylococcus epidermidis)
  4. a-hemolytic Streptococcus species (oral or viridans-group Streptococci)
  5. Corynebacterium species
  6. Candida species
  7. Enterobacterales
  8. Actinomyces species and miscellaneous aerotolerant bacteria
  9. Anaerobic bacteria with focus on Propionibacterium
Bacterial colonization 2 days after aPDT (only trauma surgery subgroup) | 2 days
  Bacterial colonization 2 days after aPDT in the midface trauma subgroup across the nine analyzed microbe groups and expressed as score (range 0-27).
  Name CFU's Score "not detectable" below detection limit 0 "sporadic" <10^4 1 "moderate" 10^4 - 10^5 2 "plentful" >10^5 3
  Nine microbial subgroups for analysis:
  1. ß-hemolytic (group A and group B) Streptococcus
  2. Staphylococcus aureus (with discrimination in MSSA and MRSA)
  3. Coagulase negative Staphylococcus species (incl. Staphylococcus epidermidis)
  4. a-hemolytic Streptococcus species (oral or viridans-group Streptococci)
  5. Corynebacterium species
  6. Candida species
  7. Enterobacterales
  8. Actinomyces species and miscellaneous aerotolerant bacteria
  9. Anaerobic bacteria with focus on Propionibacterium
Safety outcome | day 1 and day 14 (+/-1)
  Standardized survey for adverse effects noted after treatment and on day 1 and day 14 (+/-1) during regular follow-up consultation after surgery. For outpatient procedures, side effects are surveyed after treatment on the first day as a telephone conversation.

CONTACTS AND LOCATIONS:
Overall Officials: Harald Essig, Prof Dr Dr, Principal Investigator — University Hospital Zürich, Department for Oral- and Maxillofacial Surgery

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/52/NCT06570252/Prot_SAP_000.pdf